CLINICAL TRIAL: NCT06357013
Title: Postoperative Analgesia in Bilateral Knee Arthroplasties:Suprainguinal Fascia Iliaca Compartment Block and Local Infiltration Analgesia
Brief Title: Postoperative Analgesia in Bilateral Knee Arthroplasties
Status: Completed | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Yazici Kara, Principal Investigator, Kocaeli City Hospital
Other Study IDs: 2023-40
Record Dates: First submitted 2024-03-14; First posted 2024-04-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Knee Arthroplasty, Total; Peripheral Nerve Block; Pain, Postoperative
Keywords: pain; pain management; nerve block
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grup-1: Suprainguinal fascia iliaca compartment block
  Interventions: Procedure: Bilateral Suprainguinal fascia iliaca compartment block
- Grup-2: Local infiltration analgesia
  Interventions: Procedure: Local infiltration analgesia

INTERVENTIONS:
Procedure: Bilateral Suprainguinal fascia iliaca compartment block — Suprainguinal fascia iliaca compartment block (S-FICB) is one of the commonly used regional analgesia techniques for postoperative analgesia in lower extremity surgeries.
  Groups: Grup-1: Suprainguinal fascia iliaca compartment block
Procedure: Local infiltration analgesia — Local infiltration analgesia is applied to the posterior part of the knee, including the periosteum, ligaments, muscle and/or skin area before closing the surgical field.
  Groups: Grup-2: Local infiltration analgesia

SUMMARY:
To observationally compare the analgesic efficacy of LIA and S-FICB techniques and to record the pain scores of patients who underwent bilateral knee operations in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective bilateral knee arthroplasty under spinal anesthesia
* American Society of Anesthesiologists (ASA) risk score I-II
* Patients aged 18-75 years

Exclusion Criteria:

* Those receiving general anesthesia,
* Those with epidural catheters,
* Those who refused to participate in the study,
* Those whose spinal anesthesia failed and returned to general anesthesia,
* Those with a body mass index (BMI) >30 kg/m2,
* History of chronic opioid or corticosteroid use,
* Patients with psychiatric or neurological problems that would not allow assessment of pain using a visual analog scale (VAS) will be excluded.
* In addition, patients whose surgery lasted <40 minutes or >120 minutes will also be excluded to keep the data homogeneous.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years, who planned elective bilateral knee arthroplasty under spinal anesthesia, American Society of Anesthesiologists (ASA) risk score I-II.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Suprainguinal fascia iliaca compartment block (S-FICB) produces adequate analgesic effect in knee arthroplasty. | 4 months
  The aim of this study was to observationally compare the analgesic efficacy of local infiltration analgesia (LIA) and suprainguinal fascia iliaca compartment block (S-FICB) techniques in patients who underwent bilateral knee operations. Postoperative pain follow-up of the patients will be done by recording Visual analog scales (VAS) at 4, 8, 12 and 24 hours. Additional analgesic needs and unwanted side effects will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Yazici Kara, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Turkey (Türkiye)